CLINICAL TRIAL: NCT02945917
Title: Positive End-expiratory Pressure and Esophageal Catheter Optimal Calibration Volume in ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Magni Federico (Other)
Responsible Party: Sponsor-Investigator, Magni Federico, UOC Anestesia e Rianimazione ASST Monza, San Gerardo Hospital
Organization: San Gerardo Hospital (Other)
Other Study IDs: PES
Record Dates: First submitted 2016-10-20; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of esophageal balloon catheter to estimate pleural pressure has gained renewed popularity in recent years. Indeed, measurement of transpulmonary pressure may allow a more pathophysiological-based approach to ventilator strategy in acute respiratory distress syndrome (ARDS) patients. Nevertheless, it is well known that esophageal balloon catheter derived parameters can be influenced by several patient-related or technical-related factors.

During a PEEP trial, the investigators will observe in-vivo the esophageal pressure and derived measurements obtained using different esophageal balloon calibration volumes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS with a PEEP of at least 8 cmH2O
* Fraction of inspired oxygen not higher than 80%
* Intubated and ventilated in Volume Control Ventilation mode set by the attending physician according to clinical criteria
* Need of continuous sedation through intravenous anesthetics and full neuromuscular blockade

Exclusion Criteria:

* Been pregnant or breastfeeding
* Hemodynamic instability
* Presence of tracheobronchial fistula
* Known pneumothorax
* Leak in airway circuitry
* Presence of any kind of inhalator therapy (e.g. Heliox, nitric oxide, anesthetic conserving device)
* Recent history of nasal trauma or lesion of nasal cavity
* Recent history of esophageal, gastrointestinal, ENT, thoracic or cardiac surgery (less than 2 months)
* Known or suspected esophageal varices
* Congenital, acquired or drug-induced hemostatic disorder
* Thrombocytopenia (less than 50000/mm3)
* Recent history of Traumatic Brain Injury or thoraco-abdominal trauma (less than 1 months)
* Rib or sternal fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients undergoing volume control mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
transpulmonary pressure measured estimating pleural pressure through the esophageal balloon | within 10 minutes after esophageal balloon volume changing

SECONDARY OUTCOMES:
End-expiratory lung volume | within 60 minutes after PEEP changing

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Anestesia e Rianimazione, Monza, Monza E Brianza, Italy